CLINICAL TRIAL: NCT01005238
Title: A Randomized Open Label Study Evaluating the Efficacy of Continuous Telbivudine Versus Lamivudine in Patients With HBeAg-negative Chronic Hepatitis B Who Had Previously Achieved an Undetectable Viral Load During 24 Weeks of Telbivudine Therapy
Brief Title: Telbivudine Versus Lamivudine for Maintenance Therapy of Patients With Chronic Hepatitis B and Negative HBV Viral Load After 6 Month of Treatment With Telbivudine
Acronym: SASL28
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: unsufficient patient recruitment
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SASL28
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Hepatitis, Chronic
MeSH Terms: conditions — Hepatitis, Chronic | interventions — Lamivudine; Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telbivudine (Active Comparator): patients in this arm will continue to take telbivudine
  Interventions: Drug: Telbivudine
- lamivudine (Experimental): patients in this arm will take lamivudine
  Interventions: Drug: Lamivudine

INTERVENTIONS:
Drug: Lamivudine
  Arms: lamivudine
Drug: Telbivudine
  Arms: telbivudine

SUMMARY:
The aim of this randomized clinical study is to show non-inferiority of a change of anti-viral therapy from telbivudine to lamivudine in patients who have achieved an undetectable viral load at week 24 of telbivudine therapy compared to continuous treatment with telbivudine with respect to the viral breakthrough rate at week 108 as the primary clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, > 18 (having completed their 18th birthday). There is no upper limit of age
* Documented HBeAg negative CHB
* HBsAg positive > 6 months
* HBV DNA > 2000 IU/mL
* Patient is willing and able to comply with the study drug regimen and all other study requirements.
* Written informed consent
* Anti-viral HBV treatment naïve or previous treatment with interferon-alpha or pegylated interferon-alpha stopped at least 1 month prior to screening

Exclusion Criteria:

* Decompensated liver cirrhosis according to the judgment of the local investigator
* Hepatocellular carcinoma
* History of or laboratory signs of co-infection with HIV or HCV, HDV
* Previous treatment with anti-viral drugs (previous treatment with interferon-α or pegylated interferon-α is not an exclusion criteria, but has to be stopped one month before screening)
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures or their excipients
* Any medical condition that requires frequent or prolonged use of systemic corticosteroids (inhaled, topic or intra-articular corticosteroids are allowed)
* Any medical condition requiring the chronic or prolonged use of potentially hepatotoxic drugs or nephrotoxic drugs.
* Current abuse of alcohol or illicit drugs.
* Use of other investigational drugs at the time of randomization, or within 30 days or 5 half-lives of enrollment, whichever is longer.
* Any other concurrent medical or social condition which is, in the opinion of the investigator, likely to preclude compliance with the schedule of evaluations in the protocol, or likely to confound the efficacy or safety observations of the study.
* Any of the following laboratory values during Screening:

  * Hemoglobin (HGB) <11 g/dL for men or <10 g/dL for women
  * Total WBC <3000/mm3
  * Absolute neutrophil count (ANC) <1,500.mm3
  * Platelet count <50'000/mm3
  * Serum amylase or lipase ≥ 1.5 x ULN
  * Serum albumin <3 g/dL
  * Total bilirubin > 51 μmol/L (> 3.0 mg/dL)
  * Estimated calculated serum creatinine clearance < 50 mL/min using the Cockcroft-Gault method using actual or ideal body weight whichever is less (Cockcroft and Gault 1976)
  * AFP (alpha-fetoprotein) > 100 ng/mL
  * ALT > 10x ULN
* Women who are pregnant or breastfeeding. Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-HCG) during Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-09; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the rate of viral breakthrough during treatment defined as an increase of the viral titer to > 200 IU/mL. | The primary efficacy endpoint is the rate of viral breakthrough at week 108.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Heim, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland